CLINICAL TRIAL: NCT06356155
Title: A Phase II, Open-label, Single-arm, Multi-center Study of Neoadjuvant Enfortumab Vedotin and Pembrolizumab in Cisplatin-eligible Upper Tract Urothelial Cancer (NEPTUNE)
Brief Title: Study of Neoadjuvant Enfortumab Vedotin and Pembrolizumab in Cisplatin-eligible Upper Tract Urothelial Cancer
Acronym: NEPTUNE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2023.011
Record Dates: First submitted 2024-04-03; First posted 2024-04-10 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Urothelial Carcinoma
Keywords: Neoadjuvant; cisplatin-eligible
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — enfortumab vedotin; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Therapy (Experimental): Enfortumab vedotin 1.25 mg/kg IV on Days 1 and 8 and Pembrolizumab 200 mg IV on Day 1 (every 21 days for 4 cycles)
  Definitive surgery (radical nephroureterectomy RNU or distal ureterectomy per treating urologist)
  Pembrolizumab 200 mg IV on day 1 (every 21 days for up to 13 cycles) after surgery
  Interventions: Drug: Enfortumab vedotin; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Enfortumab vedotin — 1.25 mg/kg IV
  Other Names: PADCEV-EJFV
Drug: Pembrolizumab — 200 mg IV
  Other Names: Keytruda

SUMMARY:
This trial is a multi-site, single-arm, phase 2 trial of neoadjuvant combination of enfortumab vedotin and pembrolizumab in cisplatin-eligible patients with high-grade localized/locally advanced cT1-4 N0-1 M0 upper tract urothelial cancer who are deemed eligible for curative-intent surgery (radical nephroureterectomy or distal ureterectomy) followed by adjuvant pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of high-grade upper tract (renal pelvis and/or ureter) urothelial carcinoma proven by biopsy or cytology within 60 days prior to registration with the following (cT1-4 N0-1 M0): a. Upper urinary tract mass on cross-sectional imaging or Tumor directly visualized during upper urinary tract endoscopy before referral to medical oncology. b. No regional lymph node metastasis or a single regional lymph node metastasis.
* Patients must not have any component of small cell carcinoma. Other variant histologic types are permitted provided the predominant (≥50%) subtype is urothelial carcinoma.
* Patients must be considered to be a candidate for definitive surgery (nephroureterectomy or distal ureterectomy) with curative intent by the treating urologist. Lymph node dissection is strongly encouraged but its scope and determination will be at the discretion of the treating urologist. Details of the surgery such as bladder cuff removal are left to the discretion of the treating urologist. Robotic or open approaches are allowed.
* Patients must be eligible for cisplatin. Cisplatin eligibility is defined as meeting all of the following criteria: a. Creatinine clearance ≥ 45 mL/min calculated by Cockcroft-Gault equation (using actual body weight) or measured by 24-hour urine collection. b. Absence of Grade ≥ 2 peripheral neuropathy. c. Absence of New York Heart Association Class III or higher heart failure.
* Prior local endoscopic therapy for upper tract urothelial cancer is permitted if completed at least 6 months prior to the initiation of study treatment and if all toxicities from such therapy have improved to grade 1 or resolved.
* Prior uro-oncologic history: a. History of or active non-invasive carcinoma or carcinoma in situ of the bladder/urethra or upper tract is allowed. b. Patients may have received prior intravesical chemotherapy or immunotherapy such as BCG. c. Prior neoadjuvant or adjuvant chemotherapy or antibody-drug conjugate for bladder cancer or invasive contralateral upper tract cancer is allowed but must have been completed ≥ 1 year prior to study registration.
* Patients must be age ≥ 18 on the date of registration.
* ECOG Performance Status 0-1.
* Criteria for patients with hepatitis B or C are listed below. Hepatitis B and C screening tests are not required unless there is a known history of HBV or HCV infection or as mandated by local healthy authority. Hepatitis B positive subjects • Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to enrollment. • Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention. Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening. • Participants must have completed curative anti-viral therapy at least 4 weeks prior to enrollment.
* Patients must have adequate organ and bone marrow function as defined in Table 1. Specimens must be collected within 14 business days prior to start of study enrollment.
* Women and men of reproductive potential must agree to use an effective contraceptive method during treatment and for 4 months after the last dose of study drug. See Section 16.3, Appendix 3. Men must also refrain from donating sperm during this period.
* Women of reproductive potential must have a negative pregnancy test within 14 days prior to registration and are not breastfeeding.
* Patients must not have any other medical condition(s) that make(s) their participation in the study unadvisable in the opinion of the treating oncologist.
* All patients must be informed of the investigational nature of this study. The patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity who have a legally authorized representative or caregiver and/or family member available will also be considered eligible.

Exclusion Criteria:

* Prior exposure to immune-mediated therapy, including but not limited to, other anti-cytotoxic T lymphocyte-associated protein 4 (CTLA-4), anti-PD1, anti-PD-L1, anti-PD-L2 antibodies, and therapeutic anticancer vaccines.
* Prior exposure to monomethyl auristatin E antibody-drug conjugates (MMAE ADC).
* Patient is currently on or used immunosuppressive medication within 14 days prior to the first dose of pembrolizumab. The following are exceptions to this criterion: o Intranasal, inhaled, intra-auricular, topical steroids, or local steroid injections (e.g., intra-articular injection). o Use of chronic immunosuppressive agents at baseline at doses not to exceed more than prednisone 10 mg/day or equivalent. o Steroids as premedications for hypersensitivity reactions (e.g., CT scan premedication).
* Active or prior documented autoimmune or inflammatory disorders requiring immunosuppressive therapy within 2 years prior to registration. Exceptions are well-controlled hyper/hypothyroidism, celiac disease controlled by diet alone, diabetes mellitus type 1, alopecia, psoriasis, eczema, lichen planus, vitiligo, or similar skin/mucosa conditions.
* Evidence of metastasis (N2-3 or M1) on axial imaging at baseline.
* History of invasive, node positive, or metastatic bladder cancer OR invasive contralateral upper tract cancer within 2 years prior to registration.
* Enrolled in another interventional clinical trial at the time of registration.
* Patient has another active malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 1 year. The time requirement does not apply to participants who underwent successful definitive resection of non-melanoma skin cancers, superficial bladder cancer (described above in inclusion criteria 6), in situ cervical cancer, other in situ cancers, or either clinically insignificant per the investigator (e.g., ≤Gleason 3+4) on surveillance or previously treated prostate cancer without rising PSA and no plan to treat. NOTE: Patients with prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patient has one kidney.
* Patient is pregnant or lactating.
* Has severe hypersensitivity (≥ Grade 3) to enfortumab vedotin, pembrolizumab, and/or any of its excipients.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines are live attenuated vaccines and are not allowed.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has a known history of Human Immunodeficiency Virus (HIV) infection.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has had an allogenic tissue (e.g., hematopoietic stem cell transplant HSCT)/solid organ transplant.
* Has ongoing clinically significant toxicity (Grade 2 or higher with the exception of alopecia) associated with prior treatment.
* Has known active keratitis or corneal ulcerations
* Has any of the following: a. Moderate or severe liver dysfunction (does not meet hepatic function laboratory criteria outlined in Table 1). b. Uncontrolled diabetes mellitus as deemed by Hemoglobin A1c of 8 or greater.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the combination of enfortumab vedotin and pembrolizumab as neoadjuvant therapy in cisplatin-eligible patients based off pathological response | up to 16 weeks post last neoadjuvant study drug (at time of surgery)
  This trial will estimate the efficacy of combination enfortumab vedotin and pembrolizumab given as neoadjuvant therapy in cisplatin-eligible patients with localized/locally advanced upper tract urothelial cancer (cT2-4 N0-1 M0) followed by definitive surgery. The historic pT0/Ta/Tis/T1 (termed 'response' herein) rate with definitive surgery alone for a comparable patient population (H0) is approximately 20%. This study targets an improvement of 20% in the response proportion to a target 40% response rate (H1) with the combination of enfortumab vedotin and pembrolizumab. Patients who are unable to undergo definitive surgery within 16 weeks from the last dose of neoadjuvant chemotherapy will be considered non-responders for the primary endpoint.

SECONDARY OUTCOMES:
Assess the safety and toxicity of the combination of enfortumab vedotin and pembrolizumab as neoadjuvant therapy in UTUC | up to 30 days after the last dose of study treatment
  CTCAE v5 criteria will be used to assess the safety and toxicity of combination enfortumab vedotin and pembrolizumab in eligible UTUC patients. Safety and toxicity will be reported in all patients who receive treatment with any therapy on trial. Toxicity by grade and attribution will be described using counts and proportions.
Assess whether patients who receive the combination of enfortumab vedotin and pembrolizumab as neoadjuvant therapy have increased surgical complications. | up to 12 weeks after surgery
  Surgical complications will be assessed by the Clavien-Dindo classification. Grade 1 to Grade 5 (Grade 1 being no deviation and Grade 5 being death).
Estimate secondary measures of efficacy of neoadjuvant combination enfortumab vedotin and pembrolizumab and pembrolizumab adjuvant therapy (if tolerated) in response evaluable patients with UTUC by measuring RECIST v1.1 measurable disease. | up to 2 years post surgery
  Overall response in the subset of patients with RECIST v1.1 measurable disease in response evaluable patients with UTUC who receive neoadjuvant combination enfortumab vedotin and pembrolizumab will be measured. The ORR (Overall Response Rate) will be calculated from the partial responses and complete responses in the subset of subjects with have RECIST 1.1 measurable disease at baseline.
Estimate secondary measures of efficacy of neoadjuvant combination enfortumab vedotin and pembrolizumab and pembrolizumab adjuvant therapy (if tolerated) in response evaluable patients with UTUC by measuring 2-year recurrence-free survival (RFS). | up to 2 years post surgery
  2-year recurrence-free survival (RFS) proportions and 95% confidence intervals will be estimated using Kaplan-Meier methods.
Estimate secondary measures of efficacy of neoadjuvant combination enfortumab vedotin and pembrolizumab and pembrolizumab adjuvant therapy (if tolerated) in response evaluable patients with UTUC by measuring 2-year overall survival (OS). | up to 2 years post surgery
  2-year overall survival (OS) proportions and 95% confidence intervals will be estimated using Kaplan-Meier methods.
Estimate the number of patients who are able to complete neoadjuvant combination enfortumab vedotin and pembrolizumab and safely complete definitive surgery. | up to 16 weeks post last neoadjuvant study drug
  Failure to undergo surgery at all or within 16 weeks from the last dose of neoadjuvant therapy. The number of patients and associated proportion who are unable to undergo definitive surgery within 16 weeks from last dose of neoadjuvant therapy or at all will be reported.

OTHER OUTCOMES:
Assess comprehensive profiling of tumor and host characteristics (including genomics and assessment of tumor mutational burden) as predictors of response to treatment. | up to 2 years post surgery
  Integrative Next Generation Sequencing: We plan to perform integrative Next Generation Sequencing by the Michigan Center for Translational Pathology (MCTP) including but not limited to RNA-seq, PD-L1 status by the 22C3 assay, and tumor mutational burden assessment from tissue obtained at the time of diagnosis or surgery to correlate with response to treatment. Optional tumor biopsy at recurrence may be obtained for integrative next generation sequencing
Explore circulating biomarkers as early detectors of cancer recurrence | up to 2 years post surgery
  Early detection of cancer recurrence, ResBio ctDNA will be obtained prior to starting neoadjuvant therapy (cycle 1, day 1), on the last day of neoadjuvant therapy (cycle 4, day 8), after surgery at 4-6 weeks, after surgery at 12 weeks then at 3 month intervals for 24 months (after surgery).

CONTACTS AND LOCATIONS:
Overall Officials: Irene Tsung, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No